CLINICAL TRIAL: NCT00500357
Title: A Phase 3, Open-Label, Single-Arm Trial Evaluating the Safety, Tolerability, and Immunogenicity of a Subsequent Dose of 13-valent Pneumococcal Conjugate Vaccine Administered to One Group of Individuals Who Participated in Study 6115A1-500
Brief Title: Study Evaluating a 13-valent Pneumococcal Conjugate Vaccine in Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3009
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2011-02-17 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 1 dose 13vPnC

SUMMARY:
This is a follow-up study to the core study NCT00269672 (6115A1-500). This study will further evaluate the safety, tolerability, and immunogenicity of 13-valent pneumococcal conjugate vaccine (13vPnC) when administered to subjects who have already received one dose of 13vPnC, and one dose of 23-valent pneumococcal polysaccharide vaccine (23vPS) one year later. This study will determine if a subsequent dose of 13vPnC one year later results in similar or greater immune response (body's ability to protect against disease) than that measured after the initial dose of 13vPnC.

ELIGIBILITY:
* Previous participant of study 6115A1-500 and received 13vPnC +AlPO4 / 23vPS
* Generally healthy male or female adults 65 years of age or older
* Available for the duration of the trial - approximately 1 month
* No history of severe adverse reaction associated with a vaccine

  * MMSE score less than or equal to 21 was an exclusion criteria.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (12):
- South Africa (12):
  - Bishop Lavis
  - Bloemfontein
  - Brits
  - Cape Town
  - eManzimtoti
  - Lenasia
  - Paarl
  - Parow
  - Parys
  - Pretoria
  - Scottburgh South
  - Vanderbijlpark

REFERENCES:
- [Derived] Juergens C, de Villiers PJ, Moodley K, Jayawardene D, Jansen KU, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Safety and immunogenicity of 13-valent pneumococcal conjugate vaccine formulations with and without aluminum phosphate and comparison of the formulation of choice with 23-valent pneumococcal polysaccharide vaccine in elderly adults: a randomized open-label trial. Hum Vaccin Immunother. 2014;10(5):1343-53. doi: 10.4161/hv.27998. Epub 2014 Feb 27. PMID 24576885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 915 participants were enrolled in core study NCT00269672 (6115A1-500); 914 participants received 13-valent pneumococcal conjugate vaccine plus or minus aluminum phosphate (13vPnC+AlPO4 or 13vPnC-AlPO4) or 23-valent pneumococcal polysaccharide vaccine (23vPS) in Year 0 (Vaccination 1 [Vax 1]) followed by 13vPnC+AlPO4 or 23vPS in Year 1 (Vax 2).
Pre-assignment Details: 105 participants from the core study NCT00269672 (6115A1-500) who had received 13vPnC+AlPO4 (13vPnC) followed by 23vPS enrolled in the follow-up study NCT00500357 (6115A1-3009) 1 year after completion of the core study and received a subsequent 13vPnC dose at Year 2 (Vax 3).
Groups:
- 13vPnC (Vax 3 Follow-up / NCT00500357): Administered 13vPnC 0.5 milliliters (mL) intramuscularly (IM) at Year 0 (Vaccination 1 [Vax 1]) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Administered 13vPnC 0.5 mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Period: Overall Study
Arm/Group | 13vPnC (Vax 3 Follow-up / NCT00500357)
Started | 105
Received 13vPnC (Vax 3) | 105
Evaluable Immunogenicity Population | 98 (Administered Vax 1 and Vax 2 in study 6115A1-500; Vax 3 and at least 1 assay result in 6115A1-3009.)
Completed | 104
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC (Vax 3 Follow-up / NCT00500357): Administered 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Administered 13vPnC 0.5 mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Arm/Group | 13vPnC (Vax 3 Follow-up / NCT00500357)
Number analyzed (Participants) | 105
Age Continuous [Mean (Standard Deviation); unit: years] | 72.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 13 Serotypes 1 Month After 13vPnC / 23vPS / 13vPnC (Vaccination 3) Versus 1 Month After 13vPnC (Vaccination 1)
Description: Antibody geometric mean titers as measured by opsonophagocytic activity (OPA) assay for 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMTs are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Month 1 / Year 0 (Core study/NCT00269672), Month 1 / Year 2 (Follow-up study/NCT00500357)
Population: Evaluable Immunogenicity population includes participants from the evaluable immunogenicity population for Vax 1 and Vax 2 in the core study/NCT00269672, received 13vPnC in follow-up study/NCT00500357, and had at least 1 assay result in the follow-up study. N=number of participants with a determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC (Vax 1 Core Study/NCT00269672): 13vPnC 0.5 mL IM at Year 0 (Vax 1) in core study/NCT00269672 (6115A1-500).
- 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357): 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Administered 13vPnC 0.5mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Arm/Group | 13vPnC (Vax 1 Core Study/NCT00269672) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357)
Number analyzed (Participants) | 96 | 96
geometric mean titer
  Serotype 1 | 198 [133.7 to 293.0] | 78 [55.4 to 108.8]
  Serotype 3 | 126 [94.2 to 167.8] | 104 [81.5 to 132.5]
  Serotype 4 | 2210 [1603.5 to 3045.2] | 1254 [926.6 to 1695.7]
  Serotype 5 | 413 [278.0 to 614.9] | 170 [119.7 to 241.3]
  Serotype 6A | 4931 [3391.0 to 7170.8] | 3158 [2369.3 to 4209.7]
  Serotype 6B | 3251 [2105.0 to 5019.6] | 2440 [1753.2 to 3395.1]
  Serotype 7F | 869 [540.3 to 1398.0] | 353 [221.7 to 561.0]
  Serotype 9V | 977 [588.6 to 1620.4] | 247 [142.9 to 426.8]
  Serotype 14 | 982 [676.0 to 1425.8] | 550 [392.5 to 769.8]
  Serotype 18C | 2860 [1899.9 to 4304.6] | 1457 [1057.8 to 2008.1]
  Serotype 19A | 1141 [832.4 to 1564.3] | 431 [340.3 to 546.1]
  Serotype 19F | 1014 [654.4 to 1572.6] | 494 [341.4 to 715.5]
  Serotype 23F | 523 [315.4 to 867.7] | 661 [443.6 to 985.8]
Statistical Analysis 1: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 1: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — Non-inferiority declared if the lower limit of the 95 %confidence interval for the back-transformed GMFR was > 0.5 (2-fold criterion as a basis for comparison); geometric mean fold rise = 0.4, 95% CI 2-sided [0.28 to 0.56] — Confidence Intervals (CI) for the GMFR was a back transformation of a CI based on the Student t distribution for the mean difference of the logarithms of titers (Vax 3 minus [-] Vax 1)
Statistical Analysis 2: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 3: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.67 to 1.01] — CI for the GMFR was a back transformation of a CI based on the Student t distribution for the mean difference of the logarithms of titers (Vax 3 - Vax 1)
Statistical Analysis 3: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 4: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.6, 95% CI 2-sided [0.44 to 0.72] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 5: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.4, 95% CI 2-sided [0.32 to 0.53] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6A: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.6, 95% CI 2-sided [0.45 to 0.91] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6B: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.56 to 1.01] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 7F: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.4, 95% CI 2-sided [0.25 to 0.65] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 9V: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.3, 95% CI 2-sided [0.16 to 0.40] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 14: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.6, 95% CI 2-sided [0.40 to 0.78] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 18C: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.5, 95% CI 2-sided [0.40 to 0.65] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19A: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.4, 95% CI 2-sided [0.30 to 0.48] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19F: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.5, 95% CI 2-sided [0.35 to 0.67] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 23F: Geometric mean fold rise (GMFR) was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 1.3, 95% CI 2-sided [0.86 to 1.86] — [estimate comment as in outcome 1, analysis 2]

2. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination 13vPnC / 23vPS / 13vPnC (Vaccination 3)
Description: Local reactions reported using electronic diary. Redness and swelling scaled as Any (redness or swelling present); Mild (2.5 centimeters [cm] to 5.0 cm); Moderate (5.1 to 10.0 cm); Severe (> 10.0 cm). Pain scaled as Any (pain present); Mild (awareness of symptom, easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating, inability to do usual activity). Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move above head, able to move above shoulder); Severe (unable to move shoulder).
Time Frame: Days 1 through 14 / Year 2 (Follow-up study/NCT00500357)
Population: Safety population included all participants who received the vaccine sequence 13vPnC / 23vPS / 13vPnC. N=number of participants with reactogenicity events (reported Yes for at least 1 day or No for all days); (n)=number of participants with known values for 13vPnC / 23vPS / 13vPnC (Vax 3). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up/NCT00500357): Administered 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Administered 13vPnC 0.5 mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Arm/Group | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up/NCT00500357)
Number analyzed (Participants) | 91
percentage of participants
  Redness: Any (n=79) | 7.6
  Redness: Mild (n=79) | 6.3
  Redness: Moderate (n=78) | 3.8
  Redness: Severe (n=78) | 0.0
  Swelling: Any (n=83) | 16.9
  Swelling: Mild (n=81) | 12.3
  Swelling: Moderate (n=81) | 8.6
  Swelling: Severe (n=78) | 0.0
  Pain: Any (n=89) | 40.4
  Pain: Mild (n=88) | 34.1
  Pain: Moderate (n=83) | 15.7
  Pain: Severe (n=78) | 0.0
  Limitation of arm movement: Any (n=80) | 11.3
  Limitation of arm movement: Mild (n=80) | 8.8
  Limitation of arm movement: Moderate (n=78) | 2.6
  Limitation of arm movement: Severe (n=79) | 1.3

3. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination 13vPnC / 23vPS / 13vPnC (Vaccination 3)
Description: Systemic events reported using electronic diary. Fever scaled as Any (≥38 degrees Celsius [C]); Mild (≥38 but <38.5 degrees C); Moderate (≥38.5 but <39 degrees C); Severe (≥39 but ≤40 degrees C); Potentially life-threatening (>40 degrees C). Other systemic events include Fatigue, Headache, Chills, Rash, Vomiting, Decreased appetite, New muscle pain, Aggravated muscle pain, New joint pain, and Aggravated joint pain.
Time Frame: Days 1 through 14 / Year 2 (Follow-up study/NCT00500357)
Population: Safety population; N=number of participants with reactogenicity events (reported Yes for at least 1 day or No for all days); (n)=number of participants with known values for 13vPnC / 23vPS / 13vPnC (Vax 3). Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up/NCT00500357)
Number analyzed (Participants) | 91
percentage of participants
  Fever: Any ≥38 degrees C (n=81) | 7.4
  Fever: Mild ≥38 but <38.5 degrees C (n=80) | 3.8
  Fever: Moderate ≥38.5 but <39 degrees C (n=78) | 2.6
  Fever: Severe ≥39 but ≤40 degrees C (n=80) | 2.5
  Potentially life-threatening >40 degrees C (n=79) | 1.3
  Fatigue (n=83) | 27.7
  Headache (n=81) | 19.8
  Chills (n=79) | 8.9
  Rash (n=78) | 2.6
  Vomiting (n=79) | 1.3
  Decreased appetite (n=82) | 18.3
  New muscle pain (n=84) | 21.4
  Aggravated muscle pain (n=80) | 12.5
  New joint pain (n=78) | 7.7
  Aggravated joint pain (n=79) | 6.3

4. Secondary Outcome: Pneumococcal OPA Geometric Mean Titers (GMTs) for the 13 Serotypes 1 Month After 13vPnC / 23vPS / 13vPnC (Vaccination 3) Versus 1 Month After 13vPnC / 23vPS (Vaccination 2)
Description: as for outcome 1
Time Frame: Month 1 / Year 1 (Core study/NCT00269672), Month 1 / Year 2 (Follow-up study/NCT00500357)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate antibody titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Groups:
- 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672): 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500).
- 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357): 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) core study/NCT00269672. Administered 13vPnC 0.5mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Arm/Group | 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357)
Number analyzed (Participants) | 97 | 97
geometric mean titer
  Serotype 1 | 184 [136.2 to 249.2] | 81 [58.3 to 112.5]
  Serotype 3 | 131 [102.2 to 168.9] | 104 [81.5 to 132.5]
  Serotype 4 | 1457 [1092.8 to 1942.2] | 1406 [1098.1 to 1799.8]
  Serotype 5 | 326 [228.4 to 464.0] | 219 [153.6 to 312.8]
  Serotype 6A | 1732 [1163.1 to 2580.0] | 3443 [2678.7 to 4425.1]
  Serotype 6B | 1862 [1333.5 to 2600.7] | 2505 [1798.8 to 3488.1]
  Serotype 7F | 1292 [925.2 to 1803.5] | 351 [224.5 to 550.1]
  Serotype 9V | 624 [371.0 to 1051.1] | 267 [153.9 to 463.0]
  Serotype 14 | 808 [599.4 to 1089.7] | 557 [399.0 to 778.9]
  Serotype 18C | 1753 [1214.9 to 2528.5] | 1452 [1049.6 to 2009.0]
  Serotype 19A | 756 [581.2 to 983.9] | 511 [408.5 to 639.1]
  Serotype 19F | 901 [689.1 to 1177.3] | 527 [369.1 to 752.7]
  Serotype 23F | 484 [323.7 to 723.6] | 731 [499.0 to 1071.9]
Statistical Analysis 1: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 1: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.4, 95% CI 2-sided [0.34 to 0.57] — CI for the GMFR was a back transformation of a CI based on the Student t distribution for the mean difference of the logarithms of titers (Vax 3 - Vax 2)
Statistical Analysis 2: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 3: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.66 to 0.95] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 4: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 1.0, 95% CI 2-sided [0.76 to 1.22] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 5: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.7, 95% CI 2-sided [0.57 to 0.80] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6A: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 2.0, 95% CI 2-sided [1.39 to 2.84] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6B: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 1.3, 95% CI 2-sided [1.11 to 1.63] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 7F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.3, 95% CI 2-sided [0.18 to 0.41] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 9V: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.4, 95% CI 2-sided [0.27 to 0.68] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 14: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.7, 95% CI 2-sided [0.57 to 0.83] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 18C: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.8, 95% CI 2-sided [0.66 to 1.03] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19A: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.7, 95% CI 2-sided [0.58 to 0.78] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 0.6, 95% CI 2-sided [0.47 to 0.73] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 23F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; geometric mean fold rise = 1.5, 95% CI 2-sided [1.18 to 1.94] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes 1 Month After 13vPnC / 23vPS / 13vPnC (Vaccination 3) Versus 1 Month After 13vPnC (Vaccination 1)
Description: Pneumococcal IgG GMCs measured as micrograms per milliliter (mcg/mL) for the 13 pneumococcal serotypes (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F). Confidence intervals (CI) for the GMCs are back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations.
Time Frame: Month 1 / Year 0 (Core study/NCT00269672), Month 1 / Year 2 (Follow-up study/NCT00500357)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean concentration (mcg/mL)
Groups:
- 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357): 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672. Administered 13vPnC 0.5mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
Arm/Group | 13vPnC (Vax 1 Core Study/NCT00269672) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357)
Number analyzed (Participants) | 98 | 98
geometric mean concentration (mcg/mL)
  Serotype 1 | 7.67 [5.48 to 10.72] | 4.99 [4.06 to 6.14]
  Serotype 3 | 2.60 [2.04 to 3.33] | 1.35 [1.12 to 1.62]
  Serotype 4 | 4.68 [3.40 to 6.43] | 2.96 [2.30 to 3.81]
  Serotype 5 | 19.51 [13.92 to 27.36] | 6.33 [5.08 to 7.90]
  Serotype 6A | 9.12 [6.70 to 12.42] | 8.22 [6.30 to 10.72]
  Serotype 6B | 13.03 [9.11 to 18.62] | 10.32 [8.10 to 13.14]
  Serotype 7F | 6.93 [5.45 to 8.81] | 5.02 [4.23 to 5.95]
  Serotype 9V | 11.56 [8.68 to 15.40] | 5.77 [4.70 to 7.09]
  Serotype 14 | 17.51 [12.70 to 24.13] | 13.34 [10.67 to 16.69]
  Serotype 18C | 20.59 [15.35 to 27.62] | 7.82 [6.39 to 9.56]
  Serotype 19A | 29.52 [22.14 to 39.36] | 17.80 [14.67 to 21.60]
  Serotype 19F | 13.39 [9.47 to 18.92] | 8.55 [6.60 to 11.07]
  Serotype 23F | 10.16 [7.06 to 14.64] | 7.73 [5.77 to 10.36]
Statistical Analysis 1: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 1: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.65, 95% CI 2-sided [0.52 to 0.82] — CI for the GMFR was a back transformation of a CI based on the Student t distribution for the mean difference of the logarithms of concentrations (Vax 3 - Vax 1)
Statistical Analysis 2: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 3: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.52, 95% CI 2-sided [0.43 to 0.62] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 4: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.63, 95% CI 2-sided [0.53 to 0.76] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 5: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.32, 95% CI 2-sided [0.27 to 0.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6A: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.90, 95% CI 2-sided [0.74 to 1.10] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6B: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.79, 95% CI 2-sided [0.63 to 0.99] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 7F: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.72, 95% CI 2-sided [0.60 to 0.87] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 9V: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.50, 95% CI 2-sided [0.42 to 0.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 14: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.76, 95% CI 2-sided [0.59 to 0.98] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 18C: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.38, 95% CI 2-sided [0.31 to 0.46] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19A: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.60, 95% CI 2-sided [0.49 to 0.74] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19F: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.64, 95% CI 2-sided [0.52 to 0.79] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC (Vax 1 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 23F: GMFR was calculated using all participants with available data from both the Vax 1 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.76, 95% CI 2-sided [0.62 to 0.93] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes 1 Month After 13vPnC / 23vPS / 13vPnC (Vaccination 3) Versus 1 Month After 13vPnC / 23vPS (Vaccination 2)
Description: as for outcome 5
Time Frame: Month 1 / Year 1 (Core study/NCT00269672), Month 1 / Year 2 (Follow-up study/NCT00500357)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean concentration (mcg/mL)
Arm/Group | 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357)
Number analyzed (Participants) | 98 | 98
geometric mean concentration (mcg/mL)
  Serotype 1 | 7.29 [5.96 to 8.93] | 4.99 [4.06 to 6.14]
  Serotype 3 | 2.46 [2.01 to 3.01] | 1.36 [1.13 to 1.64]
  Serotype 4 | 3.93 [3.03 to 5.11] | 2.96 [2.30 to 3.81]
  Serotype 5 | 9.29 [7.37 to 11.71] | 6.33 [5.08 to 7.90]
  Serotype 6A | 5.51 [4.25 to 7.15] | 8.22 [6.30 to 10.72]
  Serotype 6B | 9.67 [7.47 to 12.53] | 10.32 [8.10 to 13.14]
  Serotype 7F | 7.41 [6.07 to 9.04] | 5.02 [4.23 to 5.95]
  Serotype 9V | 9.60 [7.68 to 12.00] | 5.77 [4.70 to 7.09]
  Serotype 14 | 22.67 [17.89 to 28.72] | 13.34 [10.67 to 16.69]
  Serotype 18C | 11.66 [9.66 to 14.07] | 7.82 [6.39 to 9.56]
  Serotype 19A | 22.78 [18.47 to 28.11] | 17.80 [14.67 to 21.60]
  Serotype 19F | 15.82 [11.97 to 20.91] | 8.55 [6.60 to 11.07]
  Serotype 23F | 7.27 [5.52 to 9.57] | 7.73 [5.77 to 10.36]
Statistical Analysis 1: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 1: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.68, 95% CI 2-sided [0.60 to 0.78] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 3: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.55, 95% CI 2-sided [0.48 to 0.64] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 4: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.75, 95% CI 2-sided [0.65 to 0.87] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 5: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.68, 95% CI 2-sided [0.61 to 0.76] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6A: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.49, 95% CI 2-sided [1.27 to 1.75] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 6B: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.07, 95% CI 2-sided [0.94 to 1.21] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 7F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.68, 95% CI 2-sided [0.58 to 0.79] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 9V: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.60, 95% CI 2-sided [0.53 to 0.68] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 14: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.59, 95% CI 2-sided [0.51 to 0.67] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 18C: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.67, 95% CI 2-sided [0.60 to 0.74] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19A: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.78, 95% CI 2-sided [0.69 to 0.88] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 19F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 0.54, 95% CI 2-sided [0.47 to 0.62] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: 13vPnC / 23vPS (Vax 2 Core Study/NCT00269672) vs 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study/NCT00500357); Serotype 23F: GMFR was calculated using all participants with available data from both the Vax 2 and Vax 3 blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.06, 95% CI 2-sided [0.90 to 1.25] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline / Day 1 up to 43 days postvaccination. Local Reactions and Systemic Events assessed within 14 days of vaccination.
Description: An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Groups:
- 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study): Administered 13vPnC 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Administered 13vPnC 0.5 mL IM at Year 2 (Vax 3) in follow-up study/NCT00500357 (6115A1-3009).
  For 13vPnC / 23vPS / 13vPnC (Vax 3 follow-up study) Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=7; systematic (solicited) Any Local Reactions N=41; systematic (solicited) Any Systemic Events N=46.
- 13vPnC+AlPO4 (After Vax 1 Core Study): Administered 13vPnC+AlPO4 0.5 mL IM at Year 0 (Vax 1) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
- 13vPnC-AlPO4 (After Vax 1 Core Study): Administered 13vPnC-AlPO4 0.5 mL IM at Year 0 (Vax 1) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
- 23vPS (After Vax 1 Core Study): Administered 23vPS 0.5 mL IM at Year 0 (Vax 1) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
- 13vPnC+AlPO4/13vPnC+AlPO4 (After Vax 2 Core Study): Administered 13vPnC + AlPO4 0.5 mL IM at Year 0 (Vax 1) followed by 13vPnC+AlPO4 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
- 13vPnC+AlPO4/23vPS (After Vax 2 Core Study): Administered 13vPnC+AlPO4 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
- 13vPnC-AlPO4/23vPS (After Vax 2 Core Study): Administered 13vPnC-AlPO4 0.5 mL IM at Year 0 (Vax 1) followed by 23vPS 0.5 mL IM at Year 1 (Vax 2) in core study/NCT00269672 (6115A1-500). Events reported Day 1 up to Day 29 postvaccination.
Arm/Group | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study) | 13vPnC+AlPO4 (After Vax 1 Core Study) | 13vPnC-AlPO4 (After Vax 1 Core Study) | 23vPS (After Vax 1 Core Study) | 13vPnC+AlPO4/13vPnC+AlPO4 (After Vax 2 Core Study) | 13vPnC+AlPO4/23vPS (After Vax 2 Core Study) | 13vPnC-AlPO4/23vPS (After Vax 2 Core Study)
Serious Adverse Events (participants affected / at risk) | 2/105 | 2/308 | 4/304 | 1/302 | 3/139 | 1/128 | 1/273
Other Adverse Events (participants affected / at risk) | 46/105 | 70/308 | 58/304 | 80/302 | 26/139 | 35/128 | 76/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study) (N=105) | 13vPnC+AlPO4 (After Vax 1 Core Study) (N=308) | 13vPnC-AlPO4 (After Vax 1 Core Study) (N=304) | 23vPS (After Vax 1 Core Study) (N=302) | 13vPnC+AlPO4/13vPnC+AlPO4 (After Vax 2 Core Study) (N=139) | 13vPnC+AlPO4/23vPS (After Vax 2 Core Study) (N=128) | 13vPnC-AlPO4/23vPS (After Vax 2 Core Study) (N=273)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Bradycardia (Cardiac disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC / 23vPS / 13vPnC (Vax 3 Follow-up Study) (N=105) | 13vPnC+AlPO4 (After Vax 1 Core Study) (N=308) | 13vPnC-AlPO4 (After Vax 1 Core Study) (N=304) | 23vPS (After Vax 1 Core Study) (N=302) | 13vPnC+AlPO4/13vPnC+AlPO4 (After Vax 2 Core Study) (N=139) | 13vPnC+AlPO4/23vPS (After Vax 2 Core Study) (N=128) | 13vPnC-AlPO4/23vPS (After Vax 2 Core Study) (N=273)
Fatigue (General disorders) | 2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Drug hypersensitivity (Immune system disorders) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Gastroenteritis (Infections and infestations) | 2 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Cystitis (Infections and infestations) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Viral rhinitis (Infections and infestations) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Headache (Nervous system disorders) | 1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Redness (any) (Skin and subcutaneous tissue disorders) | 6/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Redness (mild) (Skin and subcutaneous tissue disorders) | 5/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Redness (moderate) (Skin and subcutaneous tissue disorders) | 3/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Redness (severe) (Skin and subcutaneous tissue disorders) | 0/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Swelling (any) (Skin and subcutaneous tissue disorders) | 14/83 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Swelling (mild) (Skin and subcutaneous tissue disorders) | 10/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Swelling (moderate) (Skin and subcutaneous tissue disorders) | 7/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Swelling (severe) (Skin and subcutaneous tissue disorders) | 0/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Pain (any) (Skin and subcutaneous tissue disorders) | 36/89 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Pain (mild) (Skin and subcutaneous tissue disorders) | 30/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Pain (moderate) (Skin and subcutaneous tissue disorders) | 13/83 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Pain (severe) (Skin and subcutaneous tissue disorders) | 0/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Limitation of arm movement (any) (Skin and subcutaneous tissue disorders) | 9/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Limitation of arm movement (mild) (Skin and subcutaneous tissue disorders) | 7/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Limitation of arm movement (moderate) (Skin and subcutaneous tissue disorders) | 2/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Limitation of arm movement (severe) (Skin and subcutaneous tissue disorders) | 1/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fever (any) ≥ 38 degrees Celsius (C) (General disorders) | 6/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fever (mild) ≥ 38 but <38.5 degrees C (General disorders) | 3/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fever (moderate) ≥ 38.5 but <39 degrees C (General disorders) | 2/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fever (severe) ≥ 39 but ≤40 degrees C (General disorders) | 2/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fever (potentially life-threatening) >40 degrees C (General disorders) | 1/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Fatigue (General disorders) | 23/83 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Headache (General disorders) | 16/81 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Chills (General disorders) | 7/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Rash (General disorders) | 2/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Vomiting (General disorders) | 1/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Decreased appetitie (General disorders) | 15/82 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
New muscle pain (General disorders) | 18/84 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Aggravated muscle pain (General disorders) | 10/80 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
New joint pain (General disorders) | 6/78 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Aggravated joint pain (General disorders) | 5/79 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Lymphadenitis (Blood and lymphatic system disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0/0 | 0 | 1 | 1 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0/0 | 1 | 1 | 0 | 0 | 0 | 1
Dacryoadenitis acquired (Eye disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0/0 | 0 | 1 | 3 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0/0 | 1 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0/0 | 1 | 0 | 1 | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Anal polyp (Gastrointestinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0/0 | 9 | 17 | 22 | 5 | 8 | 17
Injection site pain (General disorders) | 0/0 | 6 | 9 | 9 | 6 | 8 | 18
Injection site movement impairment (General disorders) | 0/0 | 6 | 6 | 6 | 1 | 4 | 12
Injection site erythema (General disorders) | 0/0 | 9 | 3 | 6 | 2 | 7 | 20
Injection site swelling (General disorders) | 0/0 | 6 | 4 | 3 | 1 | 9 | 19
Pyrexia (General disorders) | 0/0 | 0 | 2 | 2 | 0 | 0 | 1
Chills (General disorders) | 0/0 | 1 | 1 | 1 | 1 | 0 | 1
Injection site inflammation (General disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site joint movement impairment (General disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0/0 | 2 | 3 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0/0 | 1 | 1 | 3 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0/0 | 3 | 0 | 2 | 1 | 1 | 4
Nasopharyngitis (Infections and infestations) | 0/0 | 0 | 2 | 2 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0/0 | 0 | 0 | 4 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0/0 | 1 | 1 | 1 | 1 | 1 | 1
Rhinitis (Infections and infestations) | 0/0 | 0 | 1 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0/0 | 0 | 0 | 3 | 0 | 1 | 3
Cellulitis (Infections and infestations) | 0/0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0/0 | 1 | 0 | 1 | 0 | 2 | 1
Cystitis (Infections and infestations) | 0/0 | 2 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0/0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Viral rhinitis (Infections and infestations) | 0/0 | 0 | 0 | 1 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0/0 | 6 | 5 | 3 | 2 | 2 | 3
Gout (Metabolism and nutrition disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/0 | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/0 | 8 | 7 | 9 | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0/0 | 6 | 7 | 10 | 4 | 7 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/0 | 2 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/0 | 1 | 1 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 2 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 1 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0/0 | 11 | 17 | 16 | 6 | 9 | 12
Dizziness (Nervous system disorders) | 0/0 | 0 | 1 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0/0 | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 1 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 2 | 3 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0/0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0/0 | 1 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0/0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.